CLINICAL TRIAL: NCT06148337
Title: Evaluation of the Effects of Eggshell Membrane in Protecting Skin From Damage Caused by Environmental Challenges and Aging
Brief Title: Eggshell Membrane Beauty From Within Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ESM Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ESM-CLN#2023T01
Record Dates: First submitted 2023-11-18; First posted 2023-11-28 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Skin Elasticity; Skin Hydration; Skin Barrier to Water Loss; Fingernail Health; Hair Health

STUDY DESIGN:
Intervention Model Description: single-center, randomized, double-blind, placebo-controlled trial design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The clinical investigator, sub-investigators, study personnel (including outcomes assessor), and study participants will be blinded to treatment until completion of the study. Only the clinical supply coordinator will be aware of treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- uESM (Ovolux brand) (Experimental): This arm will receive a treatment protocol consisting of enough capsules to provide a daily dose of one 300 mg capsule of uESM.
  Interventions: Dietary Supplement: unhydrolyzed eggshell membrane
- Placebo (Placebo Comparator): This arm will receive a treatment protocol consisting of enough capsules to provide a daily dose of one capsule containing psyllium husk fiber.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: unhydrolyzed eggshell membrane — an unhydrolyzed, minimally processed chicken eggshell membrane powder.
  Other Names: uESM; Ovolux™ brand
  Arms: uESM (Ovolux brand)
Dietary Supplement: Placebo — psyllium husk fiber powder
  Other Names: psyllium husk fiber
  Arms: Placebo

SUMMARY:
This study is intended to evaluate the efficacy of oral supplementation of an unhydrolyzed eggshell membrane ingredient (uESM) vs placebo on both objective and subjective markers of skin aging in middle-aged and senior adults using the Cutometer® MPA 580 multi-probe system along with specially designed subject questionnaires. Secondary objectives will be to assess the benefits of uESM on the health of hair and fingernails based on a subject questionnaire.

DETAILED DESCRIPTION:
This study will be conducted according to a single-center, randomized, double-blind, placebo-controlled trial design. The study protocol will be approved by an independent institutional review board (IRB) and patients will provide their written informed consent to participate. The nutritional ingredient used in this study will be unhydrolyzed eggshell membrane (uESM) (Ovolux™ brand) (ESM Technologies LLC, Carthage, MO. USA), an unhydrolyzed, minimally processed chicken eggshell membrane powder.

Up to 70 subjects will be evaluated in this placebo-controlled study at a single investigational site in the U.S. Subjects will be randomly divided into two groups of equal numbers. The first group will receive a treatment protocol consisting of enough capsules to provide a daily dose of one 300 mg capsule of uESM, the second group will receive enough capsules for one capsule daily dose containing psyllium husk fiber as a placebo treatment. Subjects will take the capsules with a morning meal for 12 consecutive weeks. Assessments will be performed at baseline (Day 0), at Week 6 and again at the end of the study (Week 12).

After a period of 10-30 minutes at the study facility for acclimation to the study center environment, skin elasticity, firmness, and fatigue will be measured using the Cutometer® MPA 580 multi-probe system by applying a constant negative pressure. Trans-epidermal water loss (TEWL) will be evaluated with the Cutometer® MPA 580 multi-probe system utilizing a Tewameter® probe, and changes in skin hydration will be measured with the Cutometer® MPA 580 multi-probe system utilizing a Corneometer® probe. Subjects will also be given questionnaires to evaluate subjective responses to skin look and feel and to evaluate subjects' observations regarding changes in the condition and growth of hair and fingernails.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be male or female, 35-70 years of age and have a light complexion
2. Subject should be generally healthy and free of chronic skin conditions
3. Subject must be able and willing to give informed consent
4. Subject must be available for and willing to attend all evaluation visits
5. Subject must not have used for 30 days prior to screening and be willing to discontinue use of all topical and ingested products expected to improve the health of the skin, hair, or fingernails for the duration of the study (Examples of these types of medicines are: tretinoin (Retin A®), isotretinoin (Accutane®), hyaluronic acid, collagen, topical steroids, topical antibiotics, topical retinol, topical benzoyl peroxide, topical glycolic acid, topical salicylic acid, etc.)
6. Subject must not be a current smoker and have not smoked cigarettes, cigars, a pipe, etc. for 3 months prior to screening and be willing to remain non-smoking for the duration of the study (the use of 'vape' pens is allowed)
7. Subjects participating in prior studies evaluating eggshell membrane can participate in the current study so long as they are not currently taking an eggshell membrane supplement and have not done so for 90 days prior to screening

Exclusion Criteria:

1. Subject has had Botox® or other facial injection (dermal filler) at or near the temple area within 6 months of screening
2. Subject has had facial cosmetic surgery affecting skin elasticity/flexibility (e.g. face lift, etc.)
3. Subject has undergone any medical procedure that would materially affect the appearance, texture or elasticity of skin at or near the evaluation sites (face or arm), as judged by the clinical investigator (e.g. chemical peel, laser resurfacing, dermaplaning, microdermabrasion, etc.) within 6 months prior to screening
4. Subject has a known eating disorder or any dysfunction affecting the digestive tract or the ability to digest food properly
5. Subject is taking any medication or substance known to impact gastric or intestinal motility or the body's ability to break down and utilize foods (i.e., weight loss drugs)
6. Subject has been diagnosed with or experienced within 30 days prior to screening any clinically significant confounding disease or condition that would interfere with the study evaluation, as judged by the clinical investigator (e.g. an allergic response resulting in hives or other skin manifestation, an outbreak of rosacea, a severe sunburn, eczema, psoriasis, skin cancer, etc.)
7. Subject has a known allergy to eggs or egg products. If any subject becomes sensitive during the study, they will immediately be excluded from continuing in the study

   a. Such sensitivity may be realized as a reaction to inoculations wherein the inoculate is derived from or contains egg components (i.e., influenza vaccine)
8. Subject body weight is greater than 350 pounds (159 kg)
9. Subject is involved in any other research study involving an investigational product (drug, device or biologic) or a new application of an approved product, within 30 days of baseline evaluation
10. Pregnant and breastfeeding women

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-12-27 (Actual); Primary Completion 2024-04-07 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
skin elasticity/firmness | 6 weeks or 12 weeks
  The primary endpoint will be any statistically significant improvement in skin firmness/elasticity in the anterior region of the temporal fossa of the face based upon measurements taken with the Cutometer® MPA 580 multi-probe system.

SECONDARY OUTCOMES:
skin hydration | 6 weeks or 12 weeks
  A secondary endpoint will be any statistically significant improvement in skin hydration in the anterior region of the temporal fossa of the face based upon measurements taken with the Cutometer® MPA 580 multi-probe system.
skin barrier function | 6 weeks or 12 weeks
  A secondary endpoint will be any statistically significant improvement in trans-epidermal water loss (TEWL) in the anterior region of the temporal fossa of the face based upon measurements taken with the Cutometer® MPA 580 multi-probe system.
overall skin health | 6 weeks or 12 weeks
  An additional secondary endpoint will be any statistically significant improvement in overall skin health versus the placebo group as determined via a Patient's Assessment. Scoring will be from 0 to 10 with 0 equating to poor and 10 equating to excellent. Higher scores equal a better outcome.
overall hair health | 6 weeks or 12 weeks
  An additional secondary endpoint will be any statistically significant improvement in hair health versus the placebo group as determined via a Patient's Assessment. Scoring will be from 0 to 10 with 0 equating to poor and 10 equating to excellent. Higher scores equal a better outcome.
overall fingernail health | 6 weeks or 12 weeks
  A final secondary endpoint will be any statistically significant improvement fingernail health versus the placebo group as determined via a Patient's Assessment. Scoring will be from 0 to 10 with 0 equating to poor and 10 equating to excellent. Higher scores equal a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Ruff, PhD, Principal Investigator — ESM Technologies, LLC d/b/a Stratum Nutrition
Locations (1):
- Stratum Nutrition National Avenue Clinic, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.

REFERENCES:
- [Background] Ovolux™ Brand Eggshell Membrane Reduces the Clinical Signs of Aging by Improving Skin, Hair & Fingernail Appearance, Texture, and Biomechanical Properties: A Single Center, Randomized, Double Blind, Placebo Controlled Clinical Trial. https://doi.org/10.4236/jcdsa.2024.144021